CLINICAL TRIAL: NCT04410510
Title: Study of the P2Et Extract Obtained From Caesalpinia Spinosa in the Symptomatic Treatment of Subjects With COVID-19 at the Hospital Universitario San Ignacio, Colombia.
Brief Title: P2Et Extract in the Symptomatic Treatment of Subjects With COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CS002-COVID19
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: COVID; Coronavirus Infection; SARS-CoV 2; COVID19
Keywords: Herbal Drug; P2Et; Caesalpinia spinosa; Coronavirus; COVID19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study to demonstrate the efficacy and safety of P2Et (Caesalpinia spinosa extract) treatment in patients with a clinical diagnosis of Covid-19 infection when added to standard therapy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: 100 patients will be randomized in a 1: 1 ratio (50 in each group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Lopinavir / ritonavir * Capsules 200/50 mg 400/100 mg every 12 hours for 7 to 14 days Hydroxychloroquine * Tab 200 mg Tab Load 400 mg every 12 hours the first day, follow 200 mg every 12 hours for 10 days Placebo capsule equivalent to 250mg of excipient every 12 hours for 14 days
  Interventions: Other: Placebo
- Intervention group (Experimental): Lopinavir / ritonavir * Capsules 200/50 mg 400/100 mg every 12 hours for 7 to 14 days Hydroxychloroquine * Tab 200 mg Tab Load 400 mg every 12 hours the first day, follow 200 mg every 12 hours for 10 days P2Et active extract capsule equivalent to 250mg of P2Et every 12 hours for 14 days
  Interventions: Drug: P2Et (Caesalpinia spinosa extract)

INTERVENTIONS:
Drug: P2Et (Caesalpinia spinosa extract) — P2Et active extract capsule equivalent to 250mg of P2Et every 12 hours for 14 days + Standard Care
  Arms: Intervention group
Other: Placebo — Placebo capsule equivalent to 250mg of excipients of P2Et every 12 hours for 14 days + Standard Care
  Arms: Control group

SUMMARY:
Antioxidants, and particularly polyphenols, have shown protection in respiratory pathologies, which is related to the decrease in the severity of the clinical picture and suppression of inflammation. This suppression of inflammation may be related to the inhibition of NF-kB polyphenols, where its activation is related to the stimulation of 150 stimuli including cytokines (IL-1β, IL-6, THF-α, GM-CSF, MCP-1), TLRs, among others. There may be other additional mechanisms that can help control virus-induced respiratory pathologies, among which are the regulation of reactive oxygen species (ROS) associated with tissue destruction caused by the virus and a selective antiviral action can be reported. direct.

The standardized P2Et extract obtained from C. spinosa, by the Immunobiology Group of the Pontificia Universidad Javeriana, is highly antioxidant, decreases lipid peroxidation and tissue damage and induces complete autophagy in stressed or tumor cells. The induction of a full autophagic flow could inhibit the replication of beta-coronaviruses like SARS-CoV-2. Furthermore, P2Et can decrease the factors involved in tissue damage by reducing IL-6 and decrease ILC2 cells of the lung in animals with lung metastases (unpublished data).

These antecedents suggest that the supplementation of patients with COVID-19 with the extract P2Et, could improve their general condition and decrease the inflammatory mediators and the viral load.

DETAILED DESCRIPTION:
Phytomedicines have been used in multiple pathologies such as cancer, diabetes, HIV and respiratory pathologies, in which the inflammatory component is characterized. The extracts of these phytomedicines have a high antioxidant capacity related to the fact that their constituents are compounds of the polyphenol type, and this antioxidant mechanism has been related in part to the antiviral action they present.

Particularly, in respiratory pathologies such as SARS-CoV, MERS-CoV, and Covid-19, an important inflammatory component is observed. Patients infected with COVID-19 have high amounts of IL1-, IFN-γ, IP-10, and MCP-1, which are likely to trigger the Th1 cellular response. Furthermore, patients requiring ICU admission have higher concentrations of G-CSF, IP-10, MCP-1, MIP1-, and TNF-α, suggesting that cytokine storm is associated with the severity of the clinical picture.

Antioxidants, and particularly polyphenols, have shown protection in respiratory pathologies, which is related to the decrease in the severity of the clinical picture and suppression of inflammation. This suppression of inflammation may be related to the inhibition of NF-kB polyphenols, where its activation is related to the stimulation of 150 stimuli including cytokines (IL-1β, IL-6, THF-α, GM-CSF, MCP-1), TLRs, among others. There may be other additional mechanisms that can help control virus-induced respiratory pathologies, among which are the regulation of reactive oxygen species (ROS) associated with tissue destruction caused by the virus and a selective antiviral action can be reported direct.

The standardized P2Et extract obtained from C. spinosa, by the Immunobiology Group of the Pontificia Universidad Javeriana, is highly antioxidant, decreases lipid peroxidation and tissue damage and induces complete autophagy in stressed or tumor cells. The induction of a full autophagic flow could inhibit the replication of beta-coronaviruses like SARS-CoV-2. Furthermore, P2Et can decrease the factors involved in tissue damage by reducing IL-6 and decrease ILC2 cells of the lung in animals with lung metastases (unpublished data).

These antecedents suggest that the supplementation of patients with COVID-19 with the extract P2Et, could improve their general condition and decrease the inflammatory mediators and the viral load.

The primary outcome is to evaluate the efficacy of P2Et in reducing the length of hospital stay of patients with clinical suspicion or confirmed case of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old.
* Diagnosis (suspected or confirmed) of COVID-19 infection, with In-hospital management indication according to the Colombian Consensus of care, diagnosis and management of SARS-COV-2 / COVID-19 infection in health care establishments (Trujillo, 2020). Recommendations based on expert consensus and informed by evidence and the recommendations of the Ministry of Health and Social Protection for April 2020.

All patients who enter the HUSI with a clinical diagnosis of COVID-19 are eligible to enter the study if they present at least one of the following indicators of respiratory compromise:

* Hypoxemia with supplemental oxygen requirements.
* Severe pneumonia: Suspicion of respiratory infection, failure of 1 organ,
* SaO2 ambient air <90% or respiratory rate> 30 resp / min.
* ARDS Acute Respiratory Distress Syndrome. Clinical findings, radiographic bilateral infiltrates + oxygenation deficit: Mild: 200 mmHg <PaO2 / FiO2 <300 mmHg. Moderate: 100 mmHg <PaO2 / FiO2 <200 mmHg. Serious: PaO2 / FiO2 <100 mmHg. If PaO2 not available SaO2 / FiO2.
* Sepsis: Defined as organic dysfunction and can be identified as an acute change in the SOFA scale> 2 points. Quick SOFA (qSOFA) with 2 of the following 3 clinical variables can identify seriously ill patients: Glasgow 13 or lower, a systolic pressure of 100 mmHg or lower and respiratory rate of 22 / min or higher. Organic insufficiency can manifest with the following alterations: Acute confusional state, Respiratory insufficiency, Reduction in the volume of diuresis, Tachycardia, Coagulopathy, Metabolic acidosis, Lactate elevation.
* Septic shock: arterial hypotension that persists after resuscitation volume and that requires vasopressors to maintain MAP> 65 mmHg and lactate> 2 mmol / L (18 mg / dL) in the absence of hypovolemia.

Exclusion Criteria:

* Negative laboratory diagnostic test for COVID-19, before randomization.
* Pregnancy.
* History of allergic reactions attributed to polyphenol type compounds similar to those found in green tea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of P2Et in reducing the length of hospital stay of patients with clinical suspicion or confirmed case of COVID-19 | 30 days
  Proportion of patients who reduce the time in the hospital

SECONDARY OUTCOMES:
Efficacy of P2Et in reducing the time to clinically significant improvement in patients with clinical suspicion or confirmed case of COVID-19 | 30 days
  Efficacy of P2Et in reducing the time to clinically significant improvement in patients with clinical suspicion or confirmed case of COVID-19
Proportion of patients with clinical suspicion or confirmed case of COVID-19, who achieve clinical improvement after 14 days of treatment | 30 days
  Evaluate the efficacy of P2Et in increasing the proportion of patients with clinical suspicion or confirmed case of COVID-19, who achieve clinical improvement after 14 days of treatment
Proportion of patients with clinical suspicion or confirmed case of COVID-19, who achieve clinical improvement after 28 days of treatment | 30 days
  Evaluate the efficacy of P2Et in increasing the proportion of patients with clinical suspicion or confirmed case of COVID-19, who achieve clinical improvement after 28 days of treatment
Efficacy of P2Et in reducing the proportion of hospitalized patients with clinical suspicion or confirmed case of COVID-19 who require admission to the ICU due to worsening clinical symptoms. | 30 days
  Assess the efficacy of P2Et in reducing the proportion of hospitalized patients with clinical suspicion or confirmed case of COVID-19 who require admission to the ICU due to worsening clinical symptoms.
Efficacy of P2Et in reducing the proportion of patients with clinical suspicion or confirmed case of COVID-19 who die from the disease. | 30 days
  Evaluate the efficacy of P2Et in reducing the proportion of patients with clinical suspicion or confirmed case of COVID-19 who die from the disease.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of the P2Et in patients with COVID-19 | 30 days
  Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of the P2Et in patients with COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Uruena C, Ballesteros-Ramirez R, Gomez-Cadena A, Barreto A, Prieto K, Quijano S, Aschner P, Martinez C, Zapata-Cardona MI, El-Ahanidi H, Jandus C, Florez-Alvarez L, Rugeles MT, Zapata-Builes W, Garcia AA, Fiorentino S. Randomized double-blind clinical study in patients with COVID-19 to evaluate the safety and efficacy of a phytomedicine (P2Et). Front Med (Lausanne). 2022 Sep 8;9:991873. doi: 10.3389/fmed.2022.991873. eCollection 2022. PMID 36160152